CLINICAL TRIAL: NCT00416910
Title: Treatment of Advanced Chronic Lymphocytic Leukemia (CLL) Fludarabine, Mitoxantrone and Cyclophosphamide With or Without G-CSF
Brief Title: Combination Chemotherapy With or Without G-CSF in Treating Patients With Relapsed Chronic Lymphocytic Leukemia
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: low recruitment
Sponsor: German CLL Study Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCLLSG-CLL6; CDR0000455571 (Registry Identifier: PDQ (Physician Data Query)); EU-20558; AMGEN-GCLLSG-CLL6; MEDAC-GCLLSG-CLL6
Record Dates: First submitted 2006-12-27; First posted 2006-12-28 (Estimated); Last update posted 2016-09-26 (Estimated); Status verified 2016-09

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: refractory chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; stage I chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Filgrastim; fludarabine; Cyclophosphamide; Mitoxantrone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- FCM (Active Comparator): Fludarabine i.v. (25 mg/m2/d, d1-3) Cyclophosphamide i.v. (200 mg/m2/d, d1-3) Mitoxantrone i.v. (8 mg/m2, d1) q28d, max. 6 cycles
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Mitoxantrone
- FCM + G-CSF (Experimental): Fludarabine i.v. (25 mg/m2/d, d1-3) Cyclophosphamide i.v. (200 mg/m2/d, d1-3) Mitoxantrone i.v. (8 mg/m2, d1) Filgrastim (G-CSF) s.c. (5 µg/kg/d beginning on day +6 until neutrophil recovery above 1500/µl.) q28d, max. 6 cycles
  Interventions: Biological: Filgrastim; Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Mitoxantrone

INTERVENTIONS:
Biological: Filgrastim
  Other Names: Neupogen
  Arms: FCM + G-CSF
Drug: Fludarabine
Drug: Cyclophosphamide
Drug: Mitoxantrone

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as fludarabine, mitoxantrone, and cyclophosphamide, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more cancer cells. Colony stimulating factors, such as G-CSF, may increase the number of immune cells found in bone marrow or peripheral blood and may help the immune system recover from the side effects of combination chemotherapy. It is not yet known whether giving combination chemotherapy alone is more effective than combination chemotherapy together with G-CSF in treating patients with chronic lymphocytic leukemia.

PURPOSE: This randomized phase III trial is studying giving combination chemotherapy together with G-CSF to see how well it works compared to giving combination chemotherapy alone in treating patients with relapsed stage I, stage II, stage III, or stage IV chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the rate of remission, severe infections, and side effects in patients with relapsed advanced chronic lymphocytic leukemia treated with fludarabine, mitoxantrone hydrochloride, and cyclophosphamide with vs without filgrastim.

Secondary

* Compare the overall survival, progression-free survival, and quality of remission in these patients.

OUTLINE: This is a multicenter, randomized study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive fludarabine IV on days 1-3, mitoxantrone hydrochloride IV on day 1, and cyclophosphamide IV on days 1-3.
* Arm II: Patients receive fludarabine, mitoxantrone hydrochloride, and cyclophosphamide as in arm I and filgrastim (G-CSF) beginning on day 6 and continuing until blood counts recover.

In both arms, treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 165 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Confirmed relapsed and advanced chronic lymphocytic leukemia (CLL)

  * Binet stage B or C disease with rapid disease progression, enlarged lymph nodes and organs, or severe B-symptoms
* No prior non-response to fludarabine combination therapy

PATIENT CHARACTERISTICS:

* ECOG performance status 0-3
* Life expectancy > 6 months
* No severe organ dysfunction
* No other prior or concurrent neoplasm, autoimmune hemolytic anemia, or thrombocytopenia

PRIOR CONCURRENT THERAPY:

* No more than three previous treatment regimens for CLL (fludarabine allowed)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 1999-07; Primary Completion 2003-09 (Actual); Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hallek, MD, Principal Investigator — Medizinische Universitaetsklinik I at the University of Cologne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: German CLL Study Group — http://www.dcllsg.de